CLINICAL TRIAL: NCT03631277
Title: Clinical and Radiographic Evaluation of Indirect Pulp Treatment of Young Permanent Molars Using Photo-Activated Oral Disinfection Versus Calcium Hydroxide: A Randomized Clinical Trial
Brief Title: Indirect Pulp Treatment of Young Permanent Molars Using Photo-Activated Oral Disinfection Versus Calcium Hydroxide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa aly fouad elchaghaby, Assistant Lecturer of Pediatric Dentistry and Dental public health, Faculty of Dentistry, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pulp capping
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Deep Caries
Keywords: Indirect pulp treatment; Photo-activated oral disinfection; Calcium Hydroxide
MeSH Terms: interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photo-activated oral disinfection (Experimental): photo-activated oral disinfection is an advanced technology utilizing two non-toxic components, a photo-activating liquid and a LED light source that selectively target and abolish cariogenic bacteria and periodontal pathogens
  Interventions: Device: photo-activated oral disinfection
- calcium hydroxide (Active Comparator): Calcium hydroxide is the gold standard for pulp capping, it permits reparative dentin bridge formation, maintains pulp vitality, protects the pulp against harmful stimuli and has antimicrobial effect
  Interventions: Drug: Calcium Hydroxide

INTERVENTIONS:
Device: photo-activated oral disinfection — Application of PAD solution using disposable tip with agitation of the solution for 60 seconds using a brush; Placement of the light disposable tip in center of lesion and holding it just above the surface; Activation of the red light for 60 seconds; (h)Sealing the cavity with glass ionomer and then filling with composite resin as a final restoration
  Other Names: PAD
  Arms: photo-activated oral disinfection
Drug: Calcium Hydroxide — calcium hydroxide( Dycal ® Dentsply Caulk )was applied using calcium hydroxide applicator followed by glass ionomer and then composite resin as a final restoration
  Other Names: Ca(OH)2
  Arms: calcium hydroxide

SUMMARY:
This study aimed to assess the clinical and radiographic success for photo-activated oral disinfection (PAD) and calcium hydroxide in indirect pulp treatment (IPT) of young permanent molars.

DETAILED DESCRIPTION:
Indirect pulp treatment is a procedure in which pulp exposure is prevented by preserving the carious dentin bordering the pulp and sealing the pulp with a biocompatible material. . Calcium hydroxide is the gold standard for pulp capping, it permits reparative dentin bridge formation, maintains pulp vitality, protects the pulp against harmful stimuli and has antimicrobial effect. However, several disadvantages were reported with its use over time including poor seal, lack of chemical and mechanical adhesion, poor strength, long-term solubility, enhanced degradation after acid etching and tunnel defects in the dentin bridge . The operative tradition is to remove softened dentin to eliminate infected tissue; however, it is impossible to eradicate all the micro-organisms because few will persist although all soft dentin was excavated.

Evidence suggest that for arresting caries lesions, it is not crucial to completely remove the infected dentin and that selective caries removal and composite restoration can yield better clinical results . For more conservative and effective treatment, disinfection instead of complete caries removal has been encouraged. . PAD is an advanced technology utilizing two non-toxic components, a photo-activating liquid and a LED light source that selectively target and abolish cariogenic bacteria and periodontal pathogens . The usage of PAD in caries management can eradicate residual bacteria in soft dentin, reassures rapid healing and improve the prognosis of treatment .

ELIGIBILITY:
Inclusion Criteria:

* Restorable lower first permanent molars with deep carious lesions
* Absence of clinical signs and symptoms of irreversible pulpitis, fistula, swelling in periodontal tissues or abnormal tooth mobility
* Absence of adverse radiographic findings
* Compliant patient/parent and (e) Absence of any systemic disease.

Exclusion Criteria:

• Previously restored teeth .

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
postoperative pain: verbal rating scale | 2 months
  categorical (No pain, Mild pain, Moderate, Severe, Very Severe, Worst possible pain ). Assessed by using verbal rating scale. minimum value is no pain while maximum value is worst possible pain. Higher values represent a worse outcome
postoperative pain: verbal rating scale | 6 months
  categorical (No pain, Mild pain, Moderate, Severe, Very Severe, Worst possible pain ). Assessed by using verbal rating scale. minimum value is no pain while maximum value is worst possible pain. Higher values represent a worse outcome
postoperative pain: verbal rating scale | 9 months
  categorical (No pain, Mild pain, Moderate, Severe, Very Severe, Worst possible pain ). Assessed by using verbal rating scale. minimum value is no pain while maximum value is worst possible pain. Higher values represent a worse outcome
postoperative pain: verbal rating scale | 12 months
  categorical (No pain, Mild pain, Moderate, Severe, Very Severe, Worst possible pain ). Assessed by using verbal rating scale. minimum value is no pain while maximum value is worst possible pain. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Presence or absence of pain on percussion | 2,6,9 and 12 months
  Binary outcome (Present or absent). Assessed by tapping the tooth with the back of the mirror
Swelling | 2,6,9 and 12 months
  Binary outcome (Present or absent). Assessed by visual examination by the examiner
Sinus or fistula | 2,6,9 and 12 months
  Binary outcome (Present or absent). Assessed by visual examination by the examiner
Adverse radiographic findings | 2,6,9 and 12 months
  Binary outcome (Present or absent). Assessed by Digora software
Thickness of newly formed dentin | 2,6,9 and 12 months
  using the Digora software. Unit of measurements were mm

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abd Alsamad, PHD, Study Director — Cairo University